CLINICAL TRIAL: NCT00693745
Title: NGAL Evaluation Along With B-Type Natriuretic Peptide in Acutely Decompensated HF
Brief Title: Neutrophil Gelatinase-Associated Lipcalin (NGAL) Evaluation Along With B-Type Natriuretic Peptide in Acutely Decompensated HF
Acronym: GALLANT
Status: Completed | Type: Observational
Sponsor: Abbott RDx Cardiometabolic (Other)
Responsible Party: Kyle Fortner, CRA, Biosite, Inc.
Other Study IDs: BSTE-0405
Record Dates: First submitted 2008-06-05; First posted 2008-06-09 (Estimated); Last update posted 2010-10-22 (Estimated); Status verified 2010-10

CONDITIONS: Acute Decompensated Heart Failure
Keywords: Acutely

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a multi-center prospective pilot clinical study to assess the utility of the Triage NGAL Test - alone and in conjunction with the Triage BNP test - as an aid in the early risk assessment for heart-failure-related adverse clinical outcomes (deaths, readmissions, and additional emergent outpatient visits) through Day 30 and Day 90 in patients presenting with acutely decompensated heart failure (HF). Its utility as an aid in the early risk assessment for renal dysfunction in patients with acutely decompensated heart failure undergoing treatment with IV diuretics will also be assessed.

DETAILED DESCRIPTION:
Approximately 200 adults presenting to the Emergency Department (ED) / hospital with acutely decompensated HF will be enrolled. EDTA anti-coagulated blood samples will be collected for measurement of blood NGAL levels (using the Triage NGAL Test) at the point of care in all subjects at up to 8 different time points from presentation until discharge.

The results of these NGAL assessments will be blinded to the medical team during the study and will not impact the medical management of the subject.

Blood samples for unblinded assessment of both serum creatinine (analyzed at the hospital's laboratory) and whole blood BNP (analyzed with the Triage BNP Test at the point-of-care or laboratory) will also be obtained at some of the same time points.

Dialysis, emergent outpatient visits for HF, hospitalizations and mortality will be recorded through Day 30 and Day 90. If an additional serum creatinine has been obtained as standard care near Day 30, it will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 years of age or older;
* Patients presenting to the emergency department / hospital with symptoms of new or decompensated heart failure and who will be treated with at least one dose of IV diuretic;
* Ability to draw blood samples for baseline NGAL, BNP and creatinine levels either prior to the administration of the first dose of IV diuretic or within 1 hour after the first dose of an IV diuretic
* Ability to provide written informed consent from subject or their authorized representative.

Exclusion Criteria:

* Acute myocardial infarction or active ischemia;
* Patients who are intubated or otherwise not able to communicate or comply with study assessments;
* Cardiogenic shock or any other clinical condition that would contraindicate the administration of an IV agent with potent vasodilating properties;
* Known history of marked renal insufficiency (e.g., usual serum creatinine ≥ 3.0 mg/dL), on dialysis (either acute of chronic) or in imminent need of dialysis at enrollment;
* Prisoners or other institutionalized or vulnerable individuals;
* Participation in an interventional clinical study within the previous 30 days;
* Unlikely to be willing or able to comply with study procedures, including the follow-up at 30 and 90 days .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the emergency department/hospital with symptoms of new or decompensated heart failure and who will be treated with at least one dose of diuretic.
Sampling Method: Non-Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2008-09; Primary Completion 2010-04 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Maisel, MD, Principal Investigator — UCSD, San Diego VA Hospital
Locations (5):
- United States (3):
  - San Diego Veterans Affairs Hospital, San Diego, California
  - New York Methodist Hospital, Brooklyn, New York
  - Ohio State University, Columbus, Ohio
- UMC Groningen (UMCG), Groningen, Netherlands
- University Hospital - Basel, Basel, Switzerland

REFERENCES:
- [Derived] Maisel AS, Mueller C, Fitzgerald R, Brikhan R, Hiestand BC, Iqbal N, Clopton P, van Veldhuisen DJ. Prognostic utility of plasma neutrophil gelatinase-associated lipocalin in patients with acute heart failure: the NGAL EvaLuation Along with B-type NaTriuretic Peptide in acutely decompensated heart failure (GALLANT) trial. Eur J Heart Fail. 2011 Aug;13(8):846-51. doi: 10.1093/eurjhf/hfr087. PMID 21791540